CLINICAL TRIAL: NCT03738462
Title: A Prospective, Multicenter Study to Evaluate the Conformis Hip System
Brief Title: A Study to Evaluate the Conformis Hip System
Status: Terminated | Type: Observational
Why Stopped: Decision of investigational team
Sponsor: Restor3D (Industry)
Responsible Party: Sponsor
Other Study IDs: 18-001
Record Dates: First submitted 2018-10-29; First posted 2018-11-13 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Clinical Condition Included in the Approved Indications For Use for the Conformis Hip System

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Conformis Hip System — The Conformis Hip System is an FDA cleared, uncemented, primary total hip replacement device composed of femoral and acetabular components. The system incorporates the use of a pre-operative CT scan to design patient-specific implants and instruments. Using patient imaging (CT scan), a patient-specific implant is designed that best meets the geometric and anatomic requirements of the specific patient. In addition, each Conformis Hip System device is shipped with an additional (optional) femoral stem (Cordera Femoral Stem).
  Other Names: Cordera Hip System

SUMMARY:
This is a prospective multicenter study. Subjects will be implanted with a Conformis Hip System. If the surgeon intraoperatively decides to use the Cordera femoral stem, these patients will also be enrolled in the study and tracked as a subset of the Conformis Hip System patient population.The study sites will be located in the United States. The study subjects will be followed for 10 years post implantation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical condition included in the approved Indications For Use for the Conformis Hip System and the Cordera Hip System
* Osteoarthritis, as confirmed by the investigator's assessment of disease status at screening visit that warrants a THR procedure
* Willingness to participate in the clinical study, to give informed consent, and to attend all follow-up visits
* > 18 years of age

Exclusion Criteria:

* Simultaneous bilateral procedure required
* BMI > 40
* Poorly controlled diabetes (defined as HbA1c>7 or Investigator discretion)
* Crowe classification of hip dysplasia, grades 2, 3, or 4
* Active malignancy (defined as a history of any invasive malignancy - except non-melanoma skin cancer), unless patient has been treated with curative intent and there have been no clinical signs or symptoms of the malignancy for at least 5 years
* Other lower extremity surgery planned within 1 year of consent to the affected limb Contralateral THR surgery within 3 months pre or post index surgery
* Neuromuscular conditions which prevent patient from participating in study activities
* Active local or systemic infection which precludes THR procedure
* Immunocompromised in the opinion of the Investigator
* Medically diagnosed fibromyalgia or similar conditions that might impact the patient's ability to differentiate source of pain
* Rheumatoid arthritis or other forms of inflammatory joint disease
* Loss of bone or musculature, osteonecrosis, neuromuscular or vascular compromise in the area of the joint to be operated on, to an extent that the procedure is unjustified
* Diagnosed with or receiving treatment for osteoporosis that is likely to confound results in the opinion of the Investigator
* Physical disability affecting the lumbar spine that is likely to confound results in the opinion of the Investigator
* Charcot or Paget's disease
* Inability to complete the protocol in the opinion of the clinical staff due to safety or other reasons
* Participation in another clinical study which would confound results
* Allergy to any of the implant materials

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with clinical condition included in the approved Indications For Use for the Conformis Hip System and the Cordera Hip System
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score | 2 Years
  Score 0-100 (successful result = post operative increase in Harris Hip Score of > 20 points + radiographically stable implant + no additional femoral reconstruction; < 70 = poor, 70-79 - fair, 80-89 = good, and 90-100 = excellent)

SECONDARY OUTCOMES:
Revision rates post-implantation | 10 Years
The Hip Injury and Osteoarthritis Outcome Score (HOOS) | 10 Years
  Score 0-100 for each of 5 subscales (symptoms, stiffness, pain, function, and quality of life)
Incidence of major procedure-related and device-related complications including infection rate | 10 Years
Post-operative leg length and implant placement in comparison to preoperative condition | Peri-operative
Utilization of fluoroscopy during implantation (number of times utilized; amount of times utilized) | Peri-operative
Length of procedure | Peri-operative
Length of hospital stay | Peri-operative
Blood management (transfusions) | Peri-operative

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - The Orthopedic Specialty Center of Northern California, Roseville, California
  - Denver Hip and Knee, Parker, Colorado
  - Personalized Orthopedic Research Institute, Boynton Beach, Florida
  - Orthopaedic Institute of Henderson, Henderson, Nevada
  - Tennessee Orthopaedic Alliance, Nashville, Tennessee
  - Scott Orthopedic Center, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: No